CLINICAL TRIAL: NCT03247205
Title: Feasibility of Extended Post-Acute Intervention for Hip Fracture Patients With Cognitive Limitations: Hip Fracture Exercise and Rehabilitation Post Hip Fracture Study (HipERS)
Brief Title: Hip Fracture Exercise and Rehabilitation Post Hip Fracture Study
Acronym: HipERS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding ran out and no subjects recruited.
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Ann Gruber-Baldini, Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HP-00073627
Record Dates: First submitted 2017-08-08; First posted 2017-08-11 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Hip Fractures; Cognitive Impairment
Keywords: hip fracture; cognitive impairment; physical therapy
MeSH Terms: conditions — Hip Fractures; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: All participants will receive the intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HipERS (Experimental): A trained physical therapist will visit each participant for a 1-hour session 3 times a week for the initial 2 weeks, and then 2 times a week for 4 weeks (total 14 hours over 6 weeks).
  Interventions: Behavioral: HipERS

INTERVENTIONS:
Behavioral: HipERS — This is a graduated, functionally-based exercise intervention conducted in the participant's home. The intervention incorporates verbal encouragement and positive reinforcement, role modeling, assessment of and elimination of unpleasant sensations associated with an activity, and confidence building through activity repetition. The exercise component includes 1) strengthening exercises, 2) range of motion exercises, 3) balance training, 4) functional training, such as chair rising, ambulation training, and stair climbing, 5) transfer practice, 6) adjusting walking aides, and 7) adapting and modifying environment; with a focus on lower extremity tasks in all these areas.

SUMMARY:
This pilot study will look at whether it is possible to give better physical therapy to people with cognitive limitations who have had a hip fracture.

DETAILED DESCRIPTION:
Although a small number of interventions have been found to be effective in improving mobility and functional recovery after a hip fracture, these studies have routinely excluded patients with cognitive limitations, a group with poor outcomes after hip fracture. It is estimated that 15-20% of all hip fracture patients experience cognitive limitation following surgery from previously undetected cognitive impairment, delirium, and other post-operative complications that persist following hospital discharge and those with cognitive limitations are slow to recover. Despite potential for a full recovery, many hip fracture patients with cognitive limitation may be discharged early from rehabilitation settings due to misperceptions about rehabilitation potential, or other psychological issues that limit their participation.

The innovation of this study is that it focuses on a critically vulnerable and costly group of patients (hip fracture patients with cognitive limitations) with an extended intervention that is tailored to the patient's needs and cognitive abilities. The post-rehabilitation period after hip fracture has been largely ignored and little is known about the effective strategies to help transition and maintain hip fracture patients (especially those with cognitive limitations) in the home setting. HipERS utilizes an effective approach to address for functional gains, but where limited attention has been given. It focuses on motivational and behavioral challenges in patients with cognitive limitations and their caregivers, which has been largely ignored in the hip fracture research

This study will gather information from 5 people with cognitive limitations who fractured a hip. Caregivers (family relative or non-relative, unpaid or paid, formal or informal) will also be invited to participate. Hip fracture participants will receive a home-based exercise intervention that will start after their "normal" rehabilitation is done. The function-based exercise intervention will be provided by physical therapists 2-3 times a week for 6 weeks. Additionally, the physical therapist will encourage the caregiver to motivate and actively engage the hip fracture participant in the therapist-prescribed home exercise program so that this can be maintained at the end of the 6-week intervention. The feasibility of the intervention will be based on the percentage of sessions participants complete. The information we get from this feasibility study will be used to plan a larger study.

ELIGIBILITY:
Hip Fracture Participant

Inclusion criteria:

* Hip fracture
* Age 65+ at time of fracture
* Had surgical repair for the hip fracture
* Completed usual rehabilitation
* Discharged to the community after rehabilitation ends (i.e., private home or assisted living)
* Cognitive limitation (MoCA score 18-25)

Exclusion criteria

* Pathologic fracture
* Not community-dwelling (e.g., nursing home resident) prior to fracture
* Bedbound during the 6 months prior to fracture
* Not returning to the community before 180 days post-hospital discharge (can go to assisted living)
* Not authorized by a physician to participate in an exercise or rehabilitation program prior to starting the intervention
* Gait speed of greater than 0.8 m/s (already walking well) at baseline

Caregiver Participant

Inclusion criteria:

* Identified as a caregiver (i.e., family relative or non-relative, unpaid or paid, informal or formal) who will help or supervise the hip fracture participant with ADL or IADL tasks after discharge from rehab
* Helping or supervising the hip fracture participant with one or more ADL or IADL tasks at least weekly when screened for this study OR plans to be the primary person providing care at least weekly after the hip fracture participant is discharged from rehab

Exclusion criteria:

* Not English speaking
* Living more than 40 miles from the hip fracture participant
* Unable to provide informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08 (Estimated); Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Feasibility of the Intervention | 6 weeks
  Data regarding feasibility will include numbers of participants contacted, enrolled, drop-outs/withdrawals, and completing intervention and the number of adverse events.
Feasibility of the Intervention (time) | 6 weeks
  Data regarding feasibility will include total time to implement the intervention.
Treatment Fidelity | 6 weeks
  Treatment fidelity of the intervention will include recording of adherence and logs of intervention tasks and problems regarding barriers to implementation of the intervention and open-ended interviews with caregivers about their experiences with the intervention.

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | 6 weeks
  Short Physical Performance Battery (SPPB) will be used to assess timed physical performance of balance, gait, strength, and endurance. Walking speed over 3 meters and a single timed chair rise without using arms will also be assessed.
Barthel Index for Activities of Daily Living | 6 weeks
  The Barthel Index will be rated by research staff after observing activity of daily living (ADL) performance. The Barthel Index is a measure of physical function that assesses a participant's ability for self-care. The Barthel Index consists of 14 items, each of which relates to a different functional activity. A total score of 100 indicates complete independence in self-care.
Lower Extremity Gain Scale (LEGS) | 6 weeks
  The Lower Extremity Gain Scale (LEGS) is a portable measure of gait and global balance, specially developed for older adults who have sustained a hip fracture. This performance measure determines how steady or unsteady the older adult is during a series of balance and gait tasks. The tasks are summarized to yield an 11-item balance score, an 8-item gait score, and a combined overall mobility score
Neuropsychiatric Inventory (NPI) | 6 weeks
  Behavioral and affective outcomes will be used to examine the impact of the intervention on behavioral symptoms of cognitive limitation using the Neuropsychiatric Inventory (NPI). The NPI includes items on 10 behavioral disturbances: delusions, hallucinations, dysphoria, anxiety, agitation/aggression, euphoria, disinhibition, irritability/lability, apathy, and aberrant motor activity. These are all rated by the caregiver.
Zarit Burden Interview | 6 weeks
  Caregiver burden will be assessed using the Zarit Burden Interview, a 22-item scale answered by caregivers, response options ranging from 0 (Never) to 4 (Nearly Always). Factors capture personal strain and role strain.
Instrumental Activities of Daily Living (IADLs) | 6 weeks
  Instrumental activities of daily living (IADLs) will be measured by 7 items from the Older Americans' Resources and Services (OARS) Activities of Daily Living Questionnaire.
Adverse Events | 6 weeks
  Falls and other adverse events, including hospitalization, nursing home placement, and death, will be recorded throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Gruber-Baldini, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No